CLINICAL TRIAL: NCT06319235
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Phase I/IIa Clinical Trial to Demonstrate the Safety and Efficacy of DUOFAG® in Bacterial Infection Treatment in Patients With Surgical Wounds
Brief Title: Clinical Trial to Demonstrate the Safety and Efficacy of DUOFAG®
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MB PHARMA s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUO2022_01; 2022-002412-23 (EudraCT Number)
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Surgical Site Infection; Staphylococcus Aureus Infection; Pseudomonas Aeruginosa Infection; Bacterial Infections; Surgical Wound Infection
Keywords: Phage Therapy; Staphylococcus aureus; Pseudomonas aeruginosa; Surgical site infection; Bacteriophage; Bacterial infections
MeSH Terms: conditions — Surgical Wound Infection; Staphylococcal Infections; Pseudomonas Infections; Bacterial Infections | interventions — Inosine Monophosphate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Experimental): DUOFAG® (the investigational medicinal product - IMP) will be administered twice a day for two weeks. DUOFAG® will be sprayed on the surgical wound. The phage titers of each bacteriophage in DUOFAG® is ≥ 10 000 000 PFU/mL (PFU = plaque forming units).
  Interventions: Drug: IMP
- Control arm (Placebo Comparator): Placebo (physiological saline solution - 0.9% sodium chloride solution) will be administered twice a day for two weeks. Placebo will be sprayed on the surgical wound.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMP — DUOFAG® is a phage cocktail (cutaneous liquid) manufactured by MB PHARMA s.r.o. and it contains bacteriophages active against Staphylococcus aureus and Pseudomonas aeruginosa.
  Other Names: DUOFAG®
  Arms: Investigational arm
Drug: Placebo — 0.9% Sodium Chloride Injection solution was manufactured by B. Braun Melsungen AG. Marketing authorization number assigned from the State Institute for drug control (Czech Republic): 76/847/92-B/C
  Other Names: 0.9% Sodium Chloride Injection
  Arms: Control arm

SUMMARY:
DUOFAG® is a phage cocktail containing bacteriophages active against Staphylococcus aureus and Pseudomonas aeruginosa. It is an investigational medicinal product for the treatment of surgical site infections caused by S. aureus and P. aeruginosa.

The primary objective of the study is to demonstrate the safety of DUOFAG® and the clinical and microbiological change within 10 weeks after the start of treatment or until healing.

DETAILED DESCRIPTION:
The study population will be recruited in two cohorts. The microbiological population of the wound will be evaluated to analyze the effect of the treatment. If the safety profile and treatment effect are going to be satisfactory, the recruitment will proceed with Cohort 2.

In both cohorts, the Investigational Medicinal Product (IMP) or placebo (the randomization ratio will be 1:1) will be applied twice a day for two weeks or until the commencement of healing.

Patients will receive the standard of care during the whole study duration. No concomitant treatment is planned during the treatment period.

The Adverse Events will be recorded on basis of an open interview without soliciting questions, and clinical observation. In case of occurrence of an adverse event (AE) with moderate or severe intensity possibly related to IMP, the treatment will be stopped, and the AE will be followed up until resolution.

Adverse Event descriptions, their severity (mild, moderate, or severe), duration and their perceived relationship to the study medication (probable, possible, unlikely, not related, and not sure) will be recorded.

The mLUMT (modified Leg Ulcer Measurement Tool) total score and individual item scores change since the baseline visit will be recorded.

Time from the start of the study treatment until the bacterial infection eradication - i. e. the swab sample is negative on S. aureus and/or P. aeruginosa will be recorded.

Time from the start of the study treatment until the wound is closed/healed (as assessed by investigator) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgical wound infection and/or dehiscence
* Wound infected by S. aureus and/or P. aeruginosa according to wound swab.
* Wound in the groin or any other skin fold as per Investigator's discretion.
* Signed Informed Consent Form, approved by the ethical committee and competent authority.
* The age between 18 and 75 years.
* Patients able and willing to comply with study procedures.
* There are no contraindications for planned concomitant medication.
* Persisting symptoms of bacterial infection < 3 weeks since the surgery.
* Women of childbearing potential must take highly effective contraceptive measures since the study start and one month after the treatment administration at a minimum.

Exclusion Criteria:

* History of an organ or bone marrow transplantation.
* Any autoimmune disease.
* Uncompensated diabetes mellitus, confirmed by the concentration of HbA1c >60 mmol/mol (6%).
* Systematic immunosuppressive therapy.
* Malignancy treatment <1 year before the Baseline visit.
* COVID-19 infection <3 months before the Baseline visit, any signs of post-COVID syndrome.
* Pregnancy or planning to become pregnant during the study.
* Breastfeeding.
* Participation in another clinical study.
* Hypersensitivity to the IMP or placebo.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint - Cohort 1 | 10 weeks (the maximum duration)
  The endpoint will be the frequency of all (local and systemic) reactions with suspected or confirmed relation to IMP.
Primary endpoint - pooled Cohorts 1 & 2 | 10 weeks (the maximum duration)
  Time to commencement of healing.

SECONDARY OUTCOMES:
Safety endpoints (assessed in pooled Cohorts 1 & 2) | 10 weeks (the maximum duration)
  The frequency of the following symptoms following the IMP application will be evaluated: local reactions, systemic reactions.
Microbiological endpoints (assessed in pooled Cohort 1 and Cohort 2) | 2 weeks (the maximum duration)
  Change of the microbiological profile of the wound assessed by swab.
Clinical efficacy endpoints | 10 weeks (the maximum duration)
  The mLUMT total score change since Baseline, time since the start of the study treatment until the bacterial infection eradication, time since the start of the study treatment until the granulation process in the wound has started, time since the start of the study treatment until the wound is closed as assessed by Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Staffa, prof., Principal Investigator — St. Anne's University Hospital Brno
Locations (1):
- St. Anne's University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MB PHARMA website — https://www.mbph.cz/duofag